CLINICAL TRIAL: NCT01282775
Title: Interventions to Control Obesity in Community Colleges
Brief Title: Interventions to Control Obesity in Community Colleges (CDC WAY to Health)
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: RTI International (Other)
Responsible Party: Laura Linnan, ScD, CHES / Associate Professor / Principal Investigator, UNC Chapel Hill
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 04-0509; DP000102 (Other Grant/Funding Number: Centers for Disease Control)
Record Dates: First submitted 2011-01-20; First posted 2011-01-25 (Estimated); Last update posted 2011-01-25 (Estimated); Status verified 2011-01

CONDITIONS: Overweight; Obesity
Keywords: overweight; obesity; worksite
MeSH Terms: conditions — Overweight; Obesity | interventions — Environment

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Environment / Usual Care (No Intervention)
- WEB+ Environment (Other): Web-based weight loss program (WEB) + Environment - Participants have access to a proven Web-based weight loss program with weekly lessons focused on lifestyle behavior changes
  Interventions: Behavioral: WEB + Environment
- WEB + Cash Incentive for Weight Loss (Other): Web-based Weight Loss Program + Cash Incentive for Weight Loss - participants have access to a proven web-based weight loss program plus they are paid cash based on the percent weight lost at 12 months compared to baseline.
  Interventions: Behavioral: WEB + Environment; Behavioral: WEB + Cash Incentive for Weight Loss

INTERVENTIONS:
Behavioral: WEB + Environment — Participants receive weekly lessons via the Web along with additional tools for weight loss support
  Other Names: Web-based Weight Loss Program
  Arms: WEB + Cash Incentive for Weight Loss; WEB+ Environment
Behavioral: WEB + Cash Incentive for Weight Loss — Participants are paid cash based on the percent weight lost at 3, 6, and 12 months.
  Other Names: Web-based weight loss program + Cash incentive
  Arms: WEB + Cash Incentive for Weight Loss

SUMMARY:
CDC WAY to Health is a three year, group-randomized weight loss intervention study where approximately 1020 overweight/obese employees nested within 17 community colleges are randomly assigned to receive one of three promising, state-of-the-art, theory-linked interventions: Environment/Usual Care (E); Web-based Weight Loss Program + Environment (WEB+E) or Web + Environment +Incentives (WEB+E+I). College is the unit of randomization and intervention; employee is the unit of analysis. Follow-up weigh-in assessments are conducted at 3, 6, and 12 months.

DETAILED DESCRIPTION:
Despite the fact that obesity is at epidemic proportions and costs US employers an estimated $78.5 billion annually; national data indicate that less than 25% of employers are offering disease management programs to address obesity. Effective weight loss programs that are adaptable to busy work environments and maintain employee interest are needed, but few rigorous tests of these programs have been attempted.

In collaboration with the North Carolina Community College System, NC Blue Cross Blue Shield, and the State Health Plan for Teachers and State Employees, this three year group-randomized weight loss intervention studies approximately 1020 overweight/obese employees nested within 17 community colleges. Campuses are randomly assigned to receive one of three promising, state-of-the-art, theory-linked interventions: Environment/Usual Care (E); Web-based Weight Loss Program + Environment (WEB+E) or Web + Environment +Incentives (WEB+E+I). College is the unit of randomization and intervention; employee is the unit of analysis. Follow-up weigh-in assessments are completed at 3, 6, and 12 months.

After formative research in Year 1 to adapt interventions for community college employees, the effects of these interventions are rigorously tested on 12-month weight loss (primary outcome). Most secondary outcomes (weight loss behaviors, moderate-vigorous physical activity; total calories, percent body fat, fruit/vegetable intake, absenteeism, productivity, medical expenditures, and quality of life) are assessed at baseline, 6 and 12 months; along with potential mediators/moderators of weight loss outcomes. Process tracking data measures fidelity, dose delivered/received and acceptability/satisfaction with the interventions. Extensive cost- and cost-effectiveness analysis, including return on investment, is undertaken. If proven effective, this strong partnership between community colleges, the State Health Plan, and the research team, will help guide program adoption and institutionalization/dissemination throughout the community college campus system.

ELIGIBILITY:
Inclusion Criteria:

* BMI greater than or equal to 25

Exclusion Criteria:

* Type I diabetes
* Pregnant or lactating
* Had a recent weight loss of 20 pounds or more
* Currently taking weight loss medication or unwilling to stop
* Undergone or scheduled weight loss surgery
* Experienced a malignancy requiring chemotherapy or radiation in the past five years
* No internet access
* Answered "yes" to the PAR-Q items and did not return a required physician's consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1029 (Actual)
Dates: Start 2005-09; Primary Completion 2006-11 (Actual); Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
weight change | 3, 6, and 12 months
  participants weight change will be analyzed at 12 months compared to baseline

SECONDARY OUTCOMES:
moderate vigorous physical activity | 3, 6, and 12 months
total calories | 3, 6, and 12 months
percent body fat | 3, 6, and 12 months
fruit/veg intake | 3, 6, and 12 months
absenteeism | 3, 6, and 12 months
quality of life | 3, 6, and 12 months
medical expenditures | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Laura A Linnan, ScD, CHES, Principal Investigator — UNC Chapel Hill